CLINICAL TRIAL: NCT06044415
Title: Brain Kinetics of Neurotransmission During JWH-018 Intoxication
Brief Title: Brain Activity Under the Influence of JWH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P145
Record Dates: First submitted 2023-08-25; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Neurotransmission During JWH Intoxication
MeSH Terms: interventions — 1-pentyl-3-(1-naphthoyl)indole; APP-CHMINACA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JWH-018 condition (Experimental)
  Interventions: Drug: JWH018
- Placebo condition (Placebo Comparator)
  Interventions: Other: non-active control (no substance)

INTERVENTIONS:
Drug: JWH018 — A vaporized dose of 7.5 mg of JWH-018 will be inhaled by the participants
  Other Names: synthetic cannabinoid
  Arms: JWH-018 condition
Other: non-active control (no substance) — Participants will inhale from a vaporizer with an empty chamber.
  Arms: Placebo condition

SUMMARY:
The goal of this placebo-controlled study is to learn about the neural mechanisms underlying the acute effects of the synthetical cannabinoid JWH-018 in healthy, occasional cannabis users. It aims to assess neural underpinnings of neurocognitive impairments and psychotomimetic symptoms expected during the intoxication. Neuronal changes similar to those seen in cannabis intoxication are expected, such as altered neurotransmission and loss of functional connectivity within the mesocorticolimbic circuit. MRS, fMRI and blood parameters will be used for assessment. Participants will be asked to complete cognitive tasks and subjective questionnaires related to the subjective experience of the drug.

ELIGIBILITY:
Inclusion Criteria:

* sufficient experience with cannabis
* Age between 18 and 40 years
* Free from psychotropic medication
* Good physical health
* Absence of any major medical, endocrine and neurological condition
* Normal weight, body mass index (weight/height^2) between 18 and 28 kg/m^2
* Written Informed Consent
* Good knowledge and understanding of the English language
* refrain from taking illicit psychoactive substances during the study
* willing to drink only alcohol-free liquids and no caffeinated beverages from 24 hours prior to dosing day, as well as during the study day
* Participants must be willing not to drive a traffic vehicle or to operate machines within 24 h after substance administration.

Exclusion Criteria:

* History of drug addiction
* Pregnancy or lactation or pregnancy planned during study participation
* Hypertension (diastolic > 90 mmHg; systolic > 140 mmHg)
* Current or history of psychiatric disorder (determined by the medical questionnaire and medical examination)
* Any chronic or acute medical condition
* History of cardiac dysfunctions (arrhythmia, ischemic heart disease,…)
* For women: no use of a reliable contraceptive
* Tobacco smoking (>20 per day)
* Excessive drinking (>20 alcoholic consumptions per week)
* Simultaneous participation in another clinical trial
* fMRI contraindications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Neurotransmission | up to 3.5 hours after drug administration
  neurochemical concentration of glutamate, GABA and dopamine measured with MRS and resting-state fMRI
Functional connectivity | during acute intoxication
  Functional connectivity strength as measured by resting-state fMRI

SECONDARY OUTCOMES:
false memory formation | up to 3.5 hours after intoxication
  Deese-Roediger-McDermott paradigm, true and false recognition scores are obtained and confidence ratings.
sustained attention | up to 3.5 hours after intoxication
  Psychomotor Vigilance Task: reaction time and attentional lapses are measured.
attentional salience processing | up to 3.5 hours after intoxication
  visual oddball paradigm: neural response to oddball vs standard stimuli presentation, reaction time is measured.
Subjective drug effects - drug liking | up to 3.5 hours after intoxication
  Sensitivity to Cannabis Reinforcement Questionnaire, scored on a 5 point scale (1= somewhat to 5 = extremely).
Subjective drug effects - subjective high | up to 3.5 hours after intoxication
  will be self-rated on a 10 cm visual analogue scale. Higher values mean more intense effects.
Subjective drug effects - dissociative state | up to 3.5 hours after intoxication
  Clinician Administered Dissociative States Scale rated on a 5 point scale. Higher values mean a more intense effect.
Subjective drug effects - psychedelic-like effects | up to 3.5 hours after intoxication
  Will be assessed using a 10cm Bowdles Visual Analogue Scale with 13 items. Higher values mean more intense effects.
Subjective drug effects - Altered States of Consciousness Rating Scale (5D-ASC) | up to 3.5 hours after intoxication
  as rated on 10cm Visual Analogue Scales. Higher values mean more intense effects.
Subjective drug effects - psychosis-like effects | up to 3.5 hours after intoxication
  Based on the investigator-rated semi-structured interview "Positive and negative syndrome scale - positive subscale", psychosis-like symptoms are rated between 1 (absent) and 7 (extreme).
Subjective drug effects - retrospective drug reinforcement (RDRV) | up to 3.5 hours after intoxication
  Self-rated questionnaire to assess tolerability and reinforcing properties. The subject has to score 1) the overall experience on a visual analog scale [VAS] (0 = intolerable to 100: well-tolerated), 2) the likelihood of using the drug again (0= not at all to 100= most of all), 3) how much they are willing to pay for the experience (€0 to €100) and 4) how likely they are to choose this over cannabis (0= not at all to 100= extremely).
JWH-018 kinetics | baseline & regular intervals up to 3.5 hours after intoxication
  JWH-018 concentration in serum
Metabolomics | baseline & regular intervals up to 3.5 hours after intoxication
  metabolomic concentration in serum
Inflammatory cytokines | at baseline & within 30 minutes after intoxication
  cytokines IL-6, TNF-alpha, and C-reactive protein concentration in serum

OTHER OUTCOMES:
Blinding quality | at end of each test day (day 1 and 2)
  Subjects are to be asked which condition they thought they received, as well as a Visual Analog Scale assessing how confident they are of their decision (0 = not at all confident, 100 = extremely confident).